CLINICAL TRIAL: NCT05647486
Title: Predictors of 30-day Postoperative Outcome After Elective Endovascular Abdominal Aortic Aneurysm Repair
Brief Title: Predictors of 30-day Postoperative Outcome After Elective EVAR
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: 30-day outcome, EVAR
Record Dates: First submitted 2022-11-22; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EVAR: Patients with AAA, treated electively by EVAR. The 30-day postoperative outcome after elective EVAR and the role of possible predictors among patients' baseline characteristics were assessed.
  Interventions: Other: 30-day postoperative outcome

INTERVENTIONS:
Other: 30-day postoperative outcome — The 30-day postoperative outcome after elective EVAR and the role of possible predictors among patients' baseline characteristics were assessed

SUMMARY:
This study investigated the 30-day postoperative outcome after elective EVAR and the role of possible predictors among patients' baseline characteristics

DETAILED DESCRIPTION:
The study included 322 consecutive AAA patients treated electively with EVAR from March 2016 to February 2019 at a tertiary referral center.

Early follow-up with clinical and laboratory evaluation took place at the 30rd day post-operatively. Any adverse event, such as major adverse cardiovascular events (MACE), post-implantation syndrome (PIS), acute kidney injury (AKI), and deaths of any cause were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Only patients managed with EVAR using standard bifurcated devices in elective setting were included.

Exclusion Criteria:

* Patients treated for ruptured, symptomatic, inflammatory or infectious AAA were excluded. Furthermore, any patient needing complex endovascular repair of the proximal landing zone was considered ineligible. Additional exclusion criteria were the presence of any trauma or surgery within two months before EVAR, any autoimmune or systemic inflammatory disease and any malignancy. Of note, any patient with clinical or laboratory signs of infection before the scheduled operation was not offered an EVAR until a complete resolution of the infection was confirmed via a clinical, laboratory and/or imaging evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included consecutive AAA patients treated electively by EVAR
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Number of patients with major adverse cardiovascular events | 30rd day post-operatively
  Number of participants with major adverse cardiovascular events
Number of patients with acute kidney injury | 30rd day post-operatively
  Number of participants with acute kidney injury according to the RIFLE (Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease) criteria
Number of patients with post-implantation syndrome | 30rd day post-operatively
  Number of participants with post-implantation syndrome SIRS, without any apparent sign of infection
Deaths of any cause | 30rd day post-operatively
  Number of participants who died from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, Professor, Study Chair — University of Thessaly
Locations (1):
- University Hospital of Larissa, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No